CLINICAL TRIAL: NCT01587950
Title: An Exploratory Study Investigating the Effects of a Potassium Nitrate Solution in Reducing Dentinal Hypersensitivity
Brief Title: The Effects of Potassium Nitrate in Reducing Dentinal Hypersensitivity
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: Z3770631
Record Dates: First submitted 2011-11-17; First posted 2012-04-30 (Estimated); Results first posted 2015-04-28 (Estimated); Last update posted 2015-04-28 (Estimated); Status verified 2013-03

CONDITIONS: Dentinal Hypersensitivity; Dental Pain
Keywords: dentinal sensitivity; potassium nitrate; dental pain
MeSH Terms: conditions — Toothache | interventions — potassium nitrate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Sterile water (Placebo Comparator): Participants to receive 250 microlitres (μL) of sterile water.
  Interventions: Drug: Placebo
- Potassium nitrate 5% solution (Experimental): Participants to receive 250 μL of potassium nitrate 5% solution.
  Interventions: Drug: Potassium Nitrate
- Potassium nitrate 2.5% solution (Experimental): Participants to receive 250 μL of potassium nitrate 2.5% solution.
  Interventions: Drug: Potassium Nitrate

INTERVENTIONS:
Drug: Potassium Nitrate — 250 μL of Potassium nitrate solution (either 5% or 2.5%)
  Arms: Potassium nitrate 2.5% solution; Potassium nitrate 5% solution
Drug: Placebo — Sterile Water
  Arms: Sterile water

SUMMARY:
A randomized, controlled, double blind exploratory study to explore the effects of two different potassium nitrate concentrations and water on exposed dentine in reducing dentinal hypersensitivity. Solutions will be applied for either 2, 5 or 10 minutes and assessed by visual analogue scale (VAS) scores following evaporative (air) stimulus.

ELIGIBILITY:
Inclusion Criteria:

* General Health and Oral Heath: Good general health and oral health with (in the opinion of the investigator) no clinically significant and relevant abnormalities of medical history.
* Teeth: Presence of teeth in various locations in the mouth to determine stent success. Required teeth include: at least three first molars; a maxillary incisor, cuspid and bicuspid; and a mandibular incisor, cuspid and bicuspid.
* Dental Sensitivity: a) Self-reported history of dentinal hypersensitivity lasting more than 6 months and a primary complaint of sensitive teeth. b) A minimum of three accessible teeth that can be isolated that meet all of the following criteria at the screening visit: i. Teeth showing signs of facial/cervical gingival recession and/or signs of erosion or abrasion. Study teeth must exhibit greater than or equal to 3mm recession at the facial surface midpoint. ii. Teeth must be visually stain and calculus free. iii. Teeth having a gingival index score less than or equal to 2. iv. Teeth with a clinical mobility of less than or equal to 1. v. Teeth that show signs of sensitivity, evaporative (air) sensitive teeth displaying a response of greater than or equal to 30 mm on a 100 mm visual analogue scale (VAS). c) A minimum of three eligible teeth identified at the screening visit that continue to show signs of sensitivity at the baseline assessment at treatment visit 1, evaporative (air) sensitive teeth displaying a response of greater than or equal to 30 mm on a 100 mm VAS.

Exclusion Criteria:

* Allergy/Intolerance: Known or suspected intolerance or hypersensitivity to the stent materials (or closely related compounds) or any of their stated ingredients.
* Condition of the Dentition: a) Sensitive teeth not expected to respond to treatment with an over-the-counter (OTC) dentifrice in the opinion of the investigator. b) Teeth with exposed dentine but with deep, defective or facial restorations, teeth used as abutments for fixed or removable partial dentures, teeth with full crowns, orthodontic bands, extensive caries or cracked enamel. Sensitive teeth with contributing aetiologies other than erosion, abrasion or recession of exposed dentine.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2009-02; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- University Park Research Center (UPRC), Fort Wayne, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at the clinical site.
Pre-assignment Details: Prior to efficacy assessment phase of this study, commercially available dental materials were employed to develop a dental stent in 3 participants. The dental stent design created a reservoir capable of holding the test solution at the cervical margin of a study tooth for at least 10 minutes. There was no efficacy data for this development phase.
Groups:
- Overall: There were six study treatment regimens- 5% Potassium nitrate (KNO3) 250μl applied to an individual tooth once for 2, 5 or 10 min; 2.5% KNO3 (250μl) applied to an individual tooth once for 2, 5 or 10 mins. Three reference treatment regimens were sterile water (250μl) applied to an individual tooth once for 2, 5 or 10 mins. Each participant received 9 treatment regimens over three treatment visits. Three individual teeth were treated at each treatment visit. Each treatment visit was one day in length. A washout of 4 days was given after each treatment visit. Study duration for each participant during this efficacy analysis phase was approximately 5 weeks
Period: Period 1
Arm/Group | Overall
Started | 12
Received 5% KNO3 Solution (5 Minutes) | 5
Received 5% KNO3 Solution (2 Minutes) | 3
Received Sterile Water (2 Minutes) | 2
Received 5% KNO3 Solution (10 Minutes) | 4
Received 2.5% KNO3 Solution (2 Minutes) | 4
Received 2.5% KNO3 Solution (10 Minutes) | 3
Received Sterile Water (10 Minutes) | 5
Received 2.5% KNO3 Solution (5 Minutes) | 5
Received Sterile Water (5 Minutes) | 5
Completed | 12
Not Completed | 0
Period: Washout 1
Arm/Group | Overall
Started | 12
Completed | 12
Not Completed | 0
Period: Period 2
Arm/Group | Overall
Started | 12
Received Sterile Water (2 Minutes) | 8
Received 5% KNO3 Solution (10 Minutes) | 4
Received 2.5% KNO3 Solution (5 Minutes) | 2
Received 2.5% KNO3 Solution (10 Minutes) | 6
Received 5% KNO3 Solution (2 Minutes) | 6
Received Sterile Water (5 Minutes) | 2
Received 2.5% KNO3 Solution (2 Minutes) | 4
Received Sterile Water (10 Minutes) | 2
Received 5% KNO3 Solution (5 Minutes) | 2
Completed | 12
Not Completed | 0
Period: Washout 2
Arm/Group | Overall
Started | 12
Completed | 12
Not Completed | 0
Period: Period 3
Arm/Group | Overall
Started | 12
Received 2.5% KNO3 Solution (2 Minutes) | 4
Received Sterile Water (10 Minutes) | 5
Received Sterile Water (2 Minutes) | 2
Received 5% KNO3 Solution (10 Minutes) | 4
Received Sterile Water (5 Minutes) | 5
Received 5% KNO3 Solution (5 Minutes) | 5
Received 5% KNO3 Solution (2 Minutes) | 3
Received 2.5% KNO3 Solution (10 Minutes) | 3
Received 2.5% KNO3 Solution (5 Minutes) | 5
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall: All randomized participants received all study treatments during this cross over study design.
Arm/Group | Overall
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: Years] | 39.0 (13.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 3
Region of Enrollment [Number; unit: Participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Adjusted Mean Change From Baseline in Evaporative Sensitivity Pain Response of Hypersensitive Tooth on a Visual Analogue Scale (VAS) Immediately Post Application of 5% KNO3 Solution, 2.5% KNO3 Solution and Sterile Water
Description: Response to a constant jet of air applied to a hypersensitive tooth was evaluated using a 100 millimeter (mm) VAS pain response scale. According to this analog scale, pain response for stimulated tooth ranged from 0 (no pain) to 100 (intense pain). Change from baseline in pain response was calculated using VAS score immediately post treatment.
Time Frame: Baseline, immediately post administration of treatment
Population: Intent to treat (ITT) population: All randomized subjects with at least one post baseline assessment of efficacy were included in analysis. Missing data was not imputed. Due to drop outs, there was difference in number of participant analyzed.
Measure: Mean (95% Confidence Interval); unit: Units on a scale
Groups:
- 2.5% KNO3 Solution (2 Minutes): Participants were administered with a maximum of 250μl of 2.5% KNO3 solution to a single sensitive tooth once for 2 minutes during each treatment period.
- 5% KNO3 Solution (2 Minutes): Participants were administered with a maximum of 250μl of 5% KNO3 solution to a single sensitive tooth once for 2 minutes during each treatment period.
- Sterile Water (2 Minutes): Participants were administered with a maximum of 250μl of sterile water to a single sensitive tooth once for 2 minutes during each treatment period.
- 2.5% KNO3 Solution (5 Minutes): Participants were administered with a maximum of 250μl of 2.5% KNO3 solution to a single sensitive tooth once for 5 minutes during each treatment period.
- 5% KNO3 Solution (5 Minutes): Participants were administered with a maximum of 250μl of 5% KNO3 solution to a single sensitive tooth once for 5 minutes during each treatment period.
- Sterile Water (5 Minutes): Participants were administered with a maximum of 250μl of sterile water to a single sensitive tooth once for 5 minutes during each treatment period.
- 2.5% KNO3 Solution (10 Minutes): Participants were administered with a maximum of 250μl of 2.5% KNO3 solution to a single sensitive tooth once for 10 minutes during each treatment period.
- 5% KNO3 Solution (10 Minutes): Participants were administered with a maximum of 250μl of 5% KNO3 solution to a single sensitive tooth once for 10 minutes during each treatment period.
- Sterile Water (10 Minutes): Participants were administered with a maximum of 250μl of sterile water to a single sensitive tooth once for 10 minutes during each treatment period.
Arm/Group | 2.5% KNO3 Solution (2 Minutes) | 5% KNO3 Solution (2 Minutes) | Sterile Water (2 Minutes) | 2.5% KNO3 Solution (5 Minutes) | 5% KNO3 Solution (5 Minutes) | Sterile Water (5 Minutes) | 2.5% KNO3 Solution (10 Minutes) | 5% KNO3 Solution (10 Minutes) | Sterile Water (10 Minutes)
Number analyzed (Participants) | 8 | 10 | 10 | 7 | 10 | 10 | 7 | 10 | 10
Units on a scale | -13.48 [-24.59 to -2.38] | -12.49 [-22.34 to -2.64] | -8.59 [-18.74 to 1.55] | -14.14 [-26.13 to -2.15] | -17.51 [-27.40 to -7.62] | -11.12 [-20.88 to -1.36] | -8.38 [-20.14 to 3.37] | -17.34 [-27.15 to -7.53] | -14.62 [-24.44 to -4.81]
Statistical Analysis 1: Comparison: 2.5% KNO3 Solution (2 Minutes) vs 5% KNO3 Solution (2 Minutes); Null hypothesis suggested that mean change from baseline in the evaporative sensitivity within each of the treatment was zero immediately post treatment. Statistical tests were 2-sided with a significance level of 0.05; Test type: Superiority or Other; p = 0.8918, ANCOVA; ANCOVA with factors for treatment group, application site, period and random effect for subject; Adjusted Mean Difference = -0.99, 95% CI 2-sided [-15.50 to 13.52] — Difference is first named treatment minus second named treatment such that a negative difference favors the first named treatment
Statistical Analysis 2: Comparison: 2.5% KNO3 Solution (2 Minutes) vs Sterile Water (2 Minutes); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.5183, ANCOVA; ANCOVA with factors for treatment group, application site, period and random effect for subject; Adjusted Mean Difference = -4.89, 95% CI 2-sided [-19.91 to 10.14] — Difference is first named treatment minus second named treatment such that a negative difference favours the first named treatment
Statistical Analysis 3: Comparison: 5% KNO3 Solution (2 Minutes) vs Sterile Water (2 Minutes); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.5718, ANCOVA; ANCOVA with factors for treatment group, application site, period and random effect for subject; Adjusted Mean Difference = -3.89, 95% CI 2-sided [-17.59 to 9.80] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: 2.5% KNO3 Solution (5 Minutes) vs 5% KNO3 Solution (5 Minutes); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.6591, ANCOVA; ANCOVA with factors for treatment group, application site, period and random effect for subject; Adjusted Mean Difference = 3.37, 95% CI 2-sided [-11.82 to 18.56] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: 2.5% KNO3 Solution (5 Minutes) vs Sterile Water (5 Minutes); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.6921, ANCOVA; ANCOVA with factors for treatment group, application site, period and random effect for subject; Adjusted Mean Difference = -3.02, 95% CI 2-sided [-18.17 to 12.13] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: 5% KNO3 Solution (5 Minutes) vs Sterile Water (5 Minutes); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.3513, ANCOVA; ANCOVA with factors for treatment group, application site, period and random effect for subject; Adjusted Mean Difference = -6.39, 95% CI 2-sided [-19.98 to 7.20] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: 2.5% KNO3 Solution (10 Minutes) vs 5% KNO3 Solution (10 Minutes); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.2346, ANCOVA; ANCOVA with factors for treatment group, application site, period and random effect for subject; Adjusted Mean Difference = 8.96, 95% CI 2-sided [-5.96 to 23.88] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 8: Comparison: 2.5% KNO3 Solution (10 Minutes) vs Sterile Water (10 Minutes); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.4138, ANCOVA; ANCOVA with factors for treatment group, application site, period and random effect for subject; Adjusted Mean Difference = 6.24, 95% CI 2-sided [-8.92 to 21.39] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 9: Comparison: 5% KNO3 Solution (10 Minutes) vs Sterile Water (10 Minutes); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.6931, ANCOVA; ANCOVA with factors for treatment group, application site, period and random effect for subject; Adjusted Mean Difference = -2.72, 95% CI 2-sided [-16.44 to 10.99] — [estimate comment as in outcome 1, analysis 2]

2. Primary Outcome: Adjusted Mean Change From Baseline in Evaporative Sensitivity Pain Response of Hypersensitive Tooth on a VAS, 10 Minutes Post Application of 5% KNO3 Solution, 2.5% KNO3 Solution and Sterile Water
Description: Response to a constant (duration, pressure, temperature, distance from target) jet of air applied to a hypersensitive tooth was evaluated using a 100 mm VAS pain response scale. According to this analog scale, pain response for stimulated tooth ranged from 0 (no pain) to 100 (intense pain). Change from baseline in pain response was calculated using VAS score at 10 minutes post treatment.
Time Frame: Baseline, 10 minutes post administration of treatment
Population: ITT population: All randomized subjects with at least one post baseline assessment of efficacy were included in analysis. Missing data was not imputed. Due to missing values, there were differences in number of participant analyzed per treatment group.
Measure: Mean (95% Confidence Interval); unit: Units on a scale
Groups:
- 5% KNO3 Solution (2 Minutes): Participants were administered with a maximum of 250μl of 5% KNO3 solution to a single sensitive tooth sensitive tooth once for 2 minutes during each treatment period.
Arm/Group | 2.5% KNO3 Solution (2 Minutes) | 5% KNO3 Solution (2 Minutes) | Sterile Water (2 Minutes) | 2.5% KNO3 Solution (5 Minutes) | 5% KNO3 Solution (5 Minutes) | Sterile Water (5 Minutes) | 2.5% KNO3 Solution (10 Minutes) | 5% KNO3 Solution (10 Minutes) | Sterile Water (10 Minutes)
Number analyzed (Participants) | 8 | 10 | 10 | 7 | 10 | 10 | 7 | 10 | 10
Units on a scale | -20.23 [-31.58 to -8.88] | -13.84 [-23.92 to -3.76] | -9.01 [-19.39 to 1.38] | -22.67 [-34.92 to -10.42] | -12.80 [-22.92 to -2.67] | -11.55 [-21.55 to -1.55] | -9.80 [-21.83 to 2.23] | -20.81 [-30.88 to -10.74] | -15.25 [-25.31 to -5.19]
Statistical Analysis 1: Comparison: 2.5% KNO3 Solution (2 Minutes) vs 5% KNO3 Solution (2 Minutes); Null hypothesis suggested that mean change from baseline in the evaporative sensitivity within each of the treatment was zero, 10 minutes post treatment. Statistical tests were 2-sided with a significance level of 0.05; Test type: Superiority or Other; p = 0.3867, ANCOVA; ANCOVA with factors for treatment group, application site, period and random effect for subject; Adjusted Mean Difference = -6.39, 95% CI 2-sided [-21.04 to 8.26] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: 2.5% KNO3 Solution (2 Minutes) vs Sterile Water (2 Minutes); [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.1448, ANCOVA; ANCOVA with factors for treatment group, application site, period and random effect for subject; Adjusted Mean Difference = -11.22, 95% CI 2-sided [-26.41 to 3.96] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: 5% KNO3 Solution (2 Minutes) vs Sterile Water (2 Minutes); [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.4874, ANCOVA; ANCOVA with factors for treatment group, application site, period and random effect for subject; Adjusted Mean Difference = -4.83, 95% CI 2-sided [-18.66 to 8.99] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 4: Comparison: 2.5% KNO3 Solution (5 Minutes) vs 5% KNO3 Solution (5 Minutes); Null hypothesis suggested that mean change from baseline in the evaporative sensitivity within the treatments was zero, 10 minutes post treatment. Statistical tests were 2-sided with a significance level of 0.05; Test type: Superiority or Other; p = 0.2038, ANCOVA; ANCOVA with factors for treatment group, application site, period and random effect for subject; Adjusted Mean Difference = -9.87, 95% CI 2-sided [-25.23 to 5.49] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 5: Comparison: 2.5% KNO3 Solution (5 Minutes) vs Sterile Water (5 Minutes); [analysis description as in outcome 2, analysis 4]; Test type: Superiority or Other; p = 0.1518, ANCOVA; ANCOVA with factors for treatment group, application site, period and random effect for subject; Adjusted Mean Difference = -11.12, 95% CI 2-sided [-26.43 to 4.19] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 6: Comparison: 5% KNO3 Solution (5 Minutes) vs Sterile Water (5 Minutes); [analysis description as in outcome 2, analysis 4]; Test type: Superiority or Other; p = 0.8567, ANCOVA; ANCOVA with factors for treatment group, application site, period and random effect for subject; Adjusted Mean Difference = -1.25, 95% CI 2-sided [-14.98 to 12.49] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 7: Comparison: 2.5% KNO3 Solution (10 Minutes) vs 5% KNO3 Solution (10 Minutes); Null hypothesis suggested that mean change from baseline in the evaporative sensitivity within the treatments was zero, at 10 minutes post treatment. Statistical tests were 2-sided with a significance level of 0.05; Test type: Superiority or Other; p = 0.1493, ANCOVA; ANCOVA with factors for treatment group, application site, period and random effect for subject; Adjusted Mean Difference = 11.01, 95% CI 2-sided [-4.06 to 26.08] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 8: Comparison: 2.5% KNO3 Solution (10 Minutes) vs Sterile Water (10 Minutes); [analysis description as in outcome 2, analysis 4]; Test type: Superiority or Other; p = 0.4798, ANCOVA; ANCOVA with factors for treatment group, application site, period and random effect for subject; Adjusted Mean Difference = 5.45, 95% CI 2-sided [-9.86 to 20.76] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 9: Comparison: 5% KNO3 Solution (10 Minutes) vs Sterile Water (10 Minutes); [analysis description as in outcome 2, analysis 4]; Test type: Superiority or Other; p = 0.4255, ANCOVA; ANCOVA with factors for treatment group, application site, period and random effect for subject; Adjusted Mean Difference = -5.56, 95% CI 2-sided [-19.42 to 8.29] — [estimate comment as in outcome 1, analysis 2]

3. Primary Outcome: Adjusted Mean Change From Baseline in Evaporative Sensitivity Pain Response of Hypersensitive Tooth on a VAS, 20 Minute Post Application of 5% KNO3 Solution, 2.5% KNO3 Solution and Sterile Water
Description: Response to a constant (duration, pressure, temperature, distance from target) jet of air applied to a hypersensitive tooth was evaluated using a 100 mm VAS pain response scale. According to this analog scale, pain response for stimulated tooth ranged from 0 (no pain) to 100 (intense pain). Change from baseline in pain response was calculated using VAS score at 20 minutes post treatment.
Time Frame: Baseline, 20 minutes post administration of treatment
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | 2.5% KNO3 Solution (2 Minutes) | 5% KNO3 Solution (2 Minutes) | Sterile Water (2 Minutes) | 2.5% KNO3 Solution (5 Minutes) | 5% KNO3 Solution (5 Minutes) | Sterile Water (5 Minutes) | 2.5% KNO3 Solution (10 Minutes) | 5% KNO3 Solution (10 Minutes) | Sterile Water (10 Minutes)
Number analyzed (Participants) | 8 | 10 | 10 | 7 | 10 | 10 | 7 | 10 | 10
Units on a scale | -22.54 [-33.96 to -11.12] | -20.58 [-30.88 to -10.29] | -16.22 [-26.78 to -5.67] | -22.25 [-34.52 to -9.98] | -16.57 [-26.88 to -6.26] | -18.23 [-28.46 to -8.00] | -12.21 [-24.38 to -0.05] | -19.97 [-30.33 to -9.61] | -18.90 [-29.21 to -8.59]
Statistical Analysis 1: Comparison: 2.5% KNO3 Solution (2 Minutes) vs 5% KNO3 Solution (2 Minutes); Null hypothesis suggested that mean change from baseline in the evaporative sensitivity within each of the treatment was zero, 20 minutes post treatment. Statistical tests were 2-sided with a significance level of 0.05; Test type: Superiority or Other; p = 0.7769, ANCOVA — ANCOVA with factors for treatment group, application site, period and random effect for subject; Adjusted Mean Difference = -1.96, 95% CI [-15.71 to 11.80] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: 2.5% KNO3 Solution (2 Minutes) vs Sterile Water (2 Minutes); [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.3811, ANCOVA; ANCOVA with factors for treatment group, application site, period and random effect for subject; Adjusted Mean Difference = -6.32, 95% CI 2-sided [-20.64 to 8.00] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: 5% KNO3 Solution (2 Minutes) vs Sterile Water (2 Minutes); [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.5044, ANCOVA; ANCOVA with factors for treatment group, application site, period and random effect for subject; Adjusted Mean Difference = -4.36, 95% CI [-17.35 to 8.63] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 4: Comparison: 2.5% KNO3 Solution (5 Minutes) vs 5% KNO3 Solution (5 Minutes); Null hypothesis suggested that mean change from baseline in the evaporative sensitivity within the treatments was zero, 20 minutes post treatment. Statistical tests were 2-sided with a significance level of 0.05; Test type: Superiority or Other; p = 0.4374, ANCOVA; ANCOVA with factors for treatment group, application site, period and random effect for subject; Adjusted Mean Difference = -5.68, 95% CI 2-sided [-20.20 to 8.84] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 5: Comparison: 2.5% KNO3 Solution (5 Minutes) vs Sterile Water (5 Minutes); [analysis description as in outcome 3, analysis 4]; Test type: Superiority or Other; p = 0.5796, ANCOVA; ANCOVA with factors for treatment group, application site, period and random effect for subject; Slope = -4.02, 95% CI 2-sided [-18.46 to 10.41] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 6: Comparison: 5% KNO3 Solution (5 Minutes) vs Sterile Water (5 Minutes); [analysis description as in outcome 3, analysis 4]; Test type: Superiority or Other; p = 0.7994, ANCOVA; ANCOVA with factors for treatment group, application site, period and random effect for subject; Adjusted Mean Difference = 1.66, 95% CI 2-sided [-11.32 to 14.64] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: 2.5% KNO3 Solution (10 Minutes) vs 5% KNO3 Solution (10 Minutes); [analysis description as in outcome 3, analysis 4]; Test type: Superiority or Other; p = 0.2784, ANCOVA; ANCOVA with factors for treatment group, application site, period and random effect for subject; Adjusted Mean Difference = 7.75, 95% CI 2-sided [-6.42 to 21.93] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 8: Comparison: 2.5% KNO3 Solution (10 Minutes) vs Sterile Water (10 Minutes); [analysis description as in outcome 3, analysis 4]; Test type: Superiority or Other; p = 0.3581, ANCOVA; ANCOVA with factors for treatment group, application site, period and random effect for subject; Adjusted Mean Difference = 6.68, 95% CI 2-sided [-7.75 to 21.12] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 9: Comparison: 5% KNO3 Solution (10 Minutes) vs Sterile Water (10 Minutes); [analysis description as in outcome 3, analysis 4]; Test type: Superiority or Other; p = 0.8703, ANCOVA; ANCOVA with factors for treatment group, application site, period and random effect for subject; Adjusted Mean Difference = -1.07, 95% CI 2-sided [-14.11 to 11.97] — [estimate comment as in outcome 1, analysis 2]

ADVERSE EVENTS:
Time Frame: All adverse events encountered or spontaneously reported following administration of any investigational product (including washout product), or for up to 5 days after the last administration of investigational product.
Groups:
- Overall: All participants received all study treatments during this cross over study design.
Arm/Group | Overall
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.